CLINICAL TRIAL: NCT03871322
Title: Rationale and Design of the Vitamin K2 and Vitamin D3 Intervention Trial in Children and Adolescents With the Low-energy Bone Fractures
Brief Title: The Vitamin K2 and D3 Intervention Trial in Children and Adolescents With the Low-energy Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Bialystok (Other)
Collaborators: Lomza State University of Applied Sciences (Unknown); International Science & Health Foundation (Unknown); American Medical Holdings Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MUBialystok1
Record Dates: First submitted 2019-03-07; First posted 2019-03-12 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Fracture Healing; Vitamin D3; Deficiency of Vitamin K2
Keywords: vitamin D; vitamin K2; low-energy fractures; fracture healing; children
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: a prospective, three- month, randomized, double-blind, placebo-controlled, intervention trial (RDBPC),
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo, same looking capsules
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Vitamin D group (Active Comparator): vitamin D supplementation - time to fracture healing
  Interventions: Dietary Supplement: Vitamin D supplementation
- Vitamin D and K2 group (Active Comparator): Vitamin D and K 2 supplementation - time of fracture healing
  Interventions: Dietary Supplement: Vitamin D and K2 supplementation
- Placebo group (Placebo Comparator): Placebo - time to fracture healing
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D and K2 supplementation — if supplementation of vitamin D and K2 changes the time to fracture healing
  Arms: Vitamin D and K2 group
Dietary Supplement: Vitamin D supplementation — if supplementation of vitamin D alone changes the time to fracture healing
  Arms: Vitamin D group
Dietary Supplement: Placebo — Placebo control group
  Arms: Placebo group

SUMMARY:
a prospective, three- month, randomized, double-blind, placebo-controlled, intervention trial (RDBPC), investigating the effect of vitamin K2 (menaquinone-7) and vitamin D3 on the healing process of low-energy bone fractures in children and adolescents

DETAILED DESCRIPTION:
At the admission of patients to the orthopedic outpatient clinic, presence of low- energy fractures will be established based on the anamnesis, physical examination and radiological evaluation. Tests to obtain the baseline blood levels of vitamin D3 will be performed, and only children with vitamin D3 levels lower than 30ng/ml in the blood will be included in the study. The selected population will then be randomly assigned by an independent investigator to the three study groups, receiving daily for three months identical- looking soft gel capsules (1 capsule/patient/day) containing supplements of vitamin D3 2,000 IU, 90 mcg of vitamin K2 as menaquinone-7 combined with 2,000 IU D3, and olive oil-containing placebo capsules respectively. During the 3-month follow-up visits to the outpatient orthopedic clinic, the pediatric orthopedist will examine the patient, evaluate the X-ray, and determine the progress in bone union and the range of joint motion. The patients will visit the clinic on weeks 1,2,4,6,8, and 12. The compliance taking the supplements will be assessed by registering a pill count returned by a patient during the scheduled visit. The blood samples will be collected upon admission to the study, day 0, and after the 3-month regimen. The blood samples will be collected for evaluation of bone turnover markers and the status of vitamin K and vitamin D3. The primary evaluation endpoints will include: the dynamics of fracture healing, changes in levels of osteocalcin, and vitamin K and vitamin D3 levels against the placebo group. The bone fracture healing milestones will be based on bone union defined as the absence of pain and the presence of bridging callus in three of the four cortices seen on the front rear projection and lateral radiographic views of the bone. Delayed union is defined as incomplete consolidation at 90 Days

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years
* Presence of low-energy fracture
* Vitamin D serum level <30ng/ml

Exclusion Criteria:

* Age > 18 years
* Lack of low-energy bone fracture
* Oral anticoagulants treatments, which interfere with vitamin K cycle
* Current supplementation with vitamin vitamins K2 or vitamin D3
* Osteogenesis imperfecta and other bone diseases
* Vitamin D concentration > 30ng/ml

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-12-24 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
time to bone union | 3 months
  The bone fracture healing milestones will be based on bone union defined as the absence of pain and the presence of bridging callus in three of the four cortices seen on the AnteroPosteral and lateral radiographs

SECONDARY OUTCOMES:
Vitamin D concentration changes | 3 months
  changes in vitamin D serum concentration
Vitamin K2 concentration changes | 3 months
  changes in vitamin K2 serum concentration
Changes in bone markers concentration | 3 months
  Changes in bone-specific alkaline phosphatase (BALP), N-terminal telopeptide (NTX)

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Popko, MD, PhD, Study Chair — Faculty of Health Sciences; Michał Karpinski, MD, Principal Investigator — Department of Pediatric Orthopedics and Traumatology; Tomasz Guszczyn, MD, PhD, Study Chair — Department of Pediatric Orthopedics and Traumatology; Sylwia Chojnowska, PhD, Study Chair — Faculty of Health Sciences Lomza; Katarzyna Maresz, PhD, Study Chair — International Science &Health Foundation; Vladimir Badmaev, Study Director — American Medical Holdings Inc
Locations (1):
- Department of Pediatric Orthopedics and Traumatology Medical University of Bialystok, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No